CLINICAL TRIAL: NCT01914679
Title: A Phase 2 Clinical Trial Evaluating Use of the NeuroPoint Medical Device as a Treatment for Fibromyalgia.
Brief Title: A Prospective Evaluation of RINCE to Reduce Fibromyalgia Effects - University of Michigan
Acronym: PERRFECT-UM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated the study
Sponsor: University of Michigan (Other)
Collaborators: Cerephex Corporation (Industry)
Responsible Party: Principal Investigator, Daniel Clauw, MD, Professor of Anesthesiology, University of Michigan
Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NPT-201-UM
Record Dates: First submitted 2013-07-23; First posted 2013-08-02 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Brain; Stimulation; Device; Treatment
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: All participants went through a 4 week sham period, followed by a 12 week intervention with the device.
Who Masked: Participant
Masking Description: Participants did not know when the stimulation was occurring or not.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sham followed by device (Experimental): 4 weeks of inactive (sham) RINCE therapy involving no RINCE therapy followed by 12 weeks of RINCE therapy involving 24 total treatments
  Interventions: Device: RINCE

INTERVENTIONS:
Device: RINCE — The intervention is repeat applications of RINCE therapy. The sham is created by not delivering the therapy stimulation signal.
  Other Names: RINCE therapy delivered by NeuroPoint Device

SUMMARY:
The purpose of this study is to evaluate the mechanisms of noninvasive cortical electrostimulation therapy known as "Reduced Impedance Noninvasive Cortical Electrostimulation" RINCE)in the management of fibromyalgia. Patients who meet the 1990 American College of Rheumatology criteria for fibromyalgia will receive up to 24 RINCE treatments delivered by a medical device called "NeuroPoint". Approximately 20 patients will receive a combination of active and inactive (sham) therapy treatments over a 16-week period followed by a 4 week post-treatment evaluation. Patients will also undergo three (3) functional brain imaging scans while participating in the study: the first prior to the commencement of treatment, another mid-treatment; and the third at the completion of the treatment period.

The study's primary outcome measure will be the change from baseline in self-reported 24-hour average pain intensity. The study's hypothesis is that there will be a change in pain intensity as well brain functioning. We do not expect there to be a statistically significant improvement in pain intensity due to the small sample but do expect to see statistically significant changes in cortical function as measured by EEG and fMRI

ELIGIBILITY:
Inclusion Criteria:

* Patient must provide written informed consent and privacy authorization prior to participation in the study. Patient must have the ability to read and/or follow written and oral instructions, abide by the study restrictions, and agree to return for the required assessments.
* Patient is female, 18-65 years of age (inclusive) at the time of consent.
* Patient must have a confirmed diagnosis of fibromyalgia meeting the ACR 1990 diagnostic criteria for fibromyalgia.
* Patients must have a 24-hour recall pain intensity score at both the screening and baseline visits between 40 and 90 inclusive on a 100 mm VAS scale.
* Female patient of childbearing potential must be willing to use an acceptable method of birth control for the duration of their study participation.
* Patients must be willing to refrain from all excluded therapies for the duration of the study.
* In the opinion of the Investigator, the patient is willing and able to comply with all protocol-specified requirements.
* Participants undergoing fMRI and 1H-MRS must be predominantly right handed (i.e. the subject writes with their right hand).

Exclusion Criteria:

The patient will not be eligible for enrollment if there is any history of, or in the opinion of the investigator, any of the following criteria are met:

* Patient has a current significant psychological or psychiatric disorder (e.g., severe, unstable or poorly controlled depression, severe anxiety or obsessive-compulsive disorder; history of suicide attempt within preceding 5 years or suicidal ideation within preceding 6 months; or any history of bipolar disorder, schizophrenia, schizoaffective or other psychotic disorder).
* Patient has a total Hospital and Anxiety Depression score of 11-21 for either anxiety or depression, or, based on the investigator's judgment, the patient is at risk of suicidal ideation or behavior.
* Patient is currently using prohibited medications or treatments (see Prohibited Concomitant Therapy section of protocol) including stimulants, anesthetic patches, CPAP and/or TENS therapy.
* Patient has an active diagnosis and is being treated for chronic infection or chronic condition such as lupus, rheumatoid arthritis, Parkinson's disease, multiple sclerosis, hepatitis, polio, seizures, or cancer (other than basal or squamous cell skin cancer).
* Patient has any other chronic pain condition other than fibromyalgia that, in the Investigator's opinion, would interfere with the assessment of fibromyalgia (e.g., rheumatoid arthritis, post herpetic neuralgia, pain associated with diabetic neuropathy, severe pain due to degenerative joint disease, etc.)
* Patient has history of seizure disorder, dementia or epilepsy anytime during his or her life except pediatric febrile seizures.
* Female patient who is pregnant, planning a pregnancy, or breastfeeding.
* Patient has any other disease or medical condition that, in the opinion of the investigator, would interfere with the evaluation of study device efficacy or safety, or would compromise the patient's ability to participate in or complete the study.
* Patient has a history of other cranial electrical stimulation device use, or electroconvulsive therapy.
* Patient has any metal implant, such as stents, aneurysm clips, shunts, pacemakers, defibrillators, neurostimulators or other contraindications with fMRI and 1H-MRS. Long-bone implants are not excluded.
* Any anticipated need for surgery that might confound results or interfere with patient's ability to comply with the protocol.
* Myocardial infarction during preceding 12 months, uncontrolled hypertension, active cardiac disease (American Heart Association Functional Class 2, 3 or 4 or Objective Class C or D), clinically significant cardiac rhythm or conduction abnormality, or anticipation of bypass or other cardiac surgery within the next 12 months.
* Current systemic infection (e.g., HIV, hepatitis).
* Patients receiving systemic corticosteroids (> 5 mg prednisone or equivalent per day).
* Pending or current litigation or disability claim (including Workman's Compensation). Patients currently receiving disability benefits will require medical monitor approval on a case-by-case basis.
* Patient has history of alcohol and/or drug abuse.
* Patient has participated in any investigational study within 30 days prior to Screening visit or is currently participating in another clinical trial.
* Patient has received any prior experimental treatment or therapy that, in the opinion of the medical monitor, would compromise the patient's ability to participate in the study.
* Patient is a staff member or relative of a staff member at either the investigative site or the Cerephex Corporation.
* Body Mass Index (BMI) of greater than approximately 40 kg/m2.
* Claustrophobia or any other factor sufficiently significant that it is likely to prevent successful completion of fMRI and 1H-MRS procedures.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Clauw, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham and RINCE Treatment: 4 weeks of inactive (sham) RINCE therapy involving no RINCE therapy (8 treatments), and 12 weeks of RINCE therapy (24 treatments).
  RINCE: The intervention is repeat applications of RINCE therapy. The sham is created by not delivering the therapy stimulation signal.
Period: Overall Study
Arm/Group | Sham and RINCE Treatment
Started | 17
Began 12 Week Actual RINCE Treatment | 17
Completed | 12
Not Completed | 5
Not completed — Lack of Efficacy | 1
Not completed — Sponsor terminated study | 4

BASELINE CHARACTERISTICS:
Groups:
- Sham and RINCE Treatment: 4 weeks of inactive (sham) RINCE therapy involving no RINCE therapy (8 treatments) and 12 weeks of RINCE therapy (24 treatments).
  RINCE: The intervention is repeat applications of RINCE therapy. The sham is created by not delivering the therapy stimulation signal.
Arm/Group | Sham and RINCE Treatment
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient 24-hour Recall Average Pain Intensity
Description: The units of measure represent self-reported average pain over the last 24 hours on a 0-100 pain rating scale where 0 is no pain and 100 is the worst pain imaginable.
  .
Time Frame: Assessed at Baseline (Week 1), Post-Sham (Week 5), Mid-Treatment (Week 10), Mid-Treatment (Week 14), Post-Treatment (Week 18)
Population: One participant missing from analysis at Week 14/Mid-Treatment/Visit 27 due to missed visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham and RINCE Treatment
Number analyzed (Participants) | 12
units on a scale
  Baseline (Week 1) | 66.42 (15.68)
  Post-Sham (Week 5) | 49.83 (29.46)
  Mid-Treatment (Week 10) | 37.50 (24.34)
  Mid-Treatment (Week 14): number analyzed (Participants) | 11
  Mid-Treatment (Week 14) | 32.18 (23.17)
  Post-Treatment (Week 18): number analyzed (Participants) | 11
  Post-Treatment (Week 18) | 32.58 (24.52)

2. Other Pre Specified Outcome: Change in Network Connectivity as Measured by EEG
Description: EEGs will be measured at the baseline, week 4, week 18 and week 21 visits.
Time Frame: Baseline (week 1), week 6, week 18 and week 21
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Investigate Changes in Neurocognitive Functioning Using the MASQ and MCS Assessments.
Description: The MASQ and MCS questionnaires will be administered at Baseline (week 1), week 6, week 10, week 14, week 18 and week 21.
Time Frame: Baseline and up to 21 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: fMRI Measures of Network Connectivity
Description: Subjects will undergo a neuroimaging scan at Baseline (week 1), week 6, and week 18. The scan will measure network connectivity during stimuli.
Time Frame: Baseline (week 1), week 6, and week 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sham and RINCE Treatment
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham and RINCE Treatment (N=17)
Loss of Balance Resulting in Fall (Injury, poisoning and procedural complications) | 4
Leg cramp (Musculoskeletal and connective tissue disorders) | 1
Cough/Congestion (Infections and infestations) | 9 (10)
Night Sweats (General disorders) | 1
Chest Pain (Cardiac disorders) | 1
Stomach Flu (achiness, diarrhea, nausea, vomiting) (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 1
Tinnitis (Ear and labyrinth disorders) | 1
Skin Tenderness (Skin and subcutaneous tissue disorders) | 1
Yeast Infection (Infections and infestations) | 1 (2)
Mental Fogginess (Psychiatric disorders) | 1
Food Poisoning (Gastrointestinal disorders) | 1
Sinus Infection (Infections and infestations) | 2
Migraine (General disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Itchy Ears/Throat (Infections and infestations) | 1
Sore Throat (Infections and infestations) | 2 (3)
Bad Dreams (Psychiatric disorders) | 1
Stomach Pain/Constipation (Gastrointestinal disorders) | 1
Ankle Pain (Injury, poisoning and procedural complications) | 1
Stomach Cramps (Gastrointestinal disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Difficulty Focusing Vision (Eye disorders) | 1
Shaking/Dizziness (General disorders) | 1

LIMITATIONS AND CAVEATS:
This mechanistic study wasn't powered to show statistically significant clinical improvement, even as originally planned. Sponsor terminated study early when they realized the devices were not delivering enough current to be of therapeutic benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No